CLINICAL TRIAL: NCT05939921
Title: Effects of Metformin Therapy on Pancreatic and Hepatic Fat Content Using 3.0 Tesla Magnetic Resonance Imaging Proton Density Fat Fraction Software in Patients of T2DM: Prospective Open Label Case Control 16 Weeks Proof of Concept Study
Brief Title: Effects of Metformin Therapy on Pancreatic and Hepatic Fat Content in Patients of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MET
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Type2diabetes
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): T2DM patients will be provided with metformin in a specified dose
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — T2DM patients will be provided with metformin in a specified dose

SUMMARY:
A sample size of 15 patients with T2DM visiting Fortis C DOC Hospital will be recruited with informed, written consent and will be requested to answer a validated questionnaire in a language known to them (English/Hindi). All these patients will undergo 2 weeks diet and exercise run in period using standard guidelines. Clinical details will be obtained from the case records of the patients. Anthropometry, skinfolds & blood pressure will be recorded as mentioned in previous studies from our group (see below for details)18,19. Overweight and, obesity will be defined according to predefined guidelines for Asian Indians20. Abdominal obesity is defined as waist circumference of ≥ 90 centimetres (cms) in males and ≥ 80 cms in females21. Each eligible subject will undergo ultrasonography of liver and pancreas before recruitment. Following ultrasonography, patients fulfilling the inclusion will be randomised to receive the 10 mg of Dapagliflozin as mentioned previously. Biochemistry, ultrasonography, DEXA, MRI, will be performed at baseline and at 4 months post intervention.

DETAILED DESCRIPTION:
A chronic metabolic disorder described by continuous hyperglycemia we call Diabetes mellitus or DM. this metabolic disorder could be for various reasons like resisting to marginal action of insulin, also could be due to diminished secretion of insulin, or maybe both. This Chronic hyperglycemia could be responsible for other kinds of abnormalities and therefore damage various organs in the patient, sometimes this also could even be life threatening complications.

NAFLD (Nonalcoholic fatty liver disease) has the highest incidence rate among obese and diabetic patients. In various studies, it has been found that Type 2 diabetes mellitus (T2DM) and nonalcoholic fatty liver disease (NAFLD) exist together which is a metabolic disorder. It has been found that the occurrence of NAFLD is 59.67% among T2DM patients with nonalcoholic steatohepatitis (NASH), simple steatosis (NAFL), and cirrhosis.

The studies reveal that NAFLD of 70% is usually found among T2DM patients. It is also observed that obesity and insulin resistance is correlated with NAFLD.

Noninvasive assessment and staging of disease are based on clinical parameters such as age, sex, liver function test, platelet count, lipid profile, BMI, and imaging modalities such as USG, Fibro-scan (FS), and magnetic resonance imaging mass spectroscopy. Such clinical scoring systems and TE are useful in the early detection of NAFLD and predicting fibrosis. The principle behind the management of NAFLD with T2DM involves an indirect effect through improvement in IR and glycemia and thus is used for the treatment of T2DM as well.

In addition to this, fatty pancreas is gaining importance from the research point of view. Study done by our group also showed that subcutaneous and intra-abdominal obesity, including fatty liver and pancreatic volume, were larger in non-obese Asian Indians with type 2 diabetes than in BMI-matched non-diabetic participants, whereas peripheral subcutaneous adiposity was lower. A study done in animal model shows that metformin exerted a beneficial effect in limiting beta-proliferation caused by high fat diet (HFD) fed to mice and also improved insulin resistance. Another study also showed similar effects of Metformin therapy, as it decreased the amount of fat in the liver in parallel with an improvement in the metabolic parameters and may, thus, be beneficial for preventing the late consequences of NAFLD in newly diagnosed diabetic patients.

The study mentioned below predicted that Metformin would considerably reduce pancreatic and liver fat in T2DM patients. Metformin does not appear to cause or exacerbate liver injury and, indeed, is often beneficial in patients with nonalcoholic fatty liver disease. Nonalcoholic fatty liver frequently presents with transaminase elevations but should not be considered a contraindication to metformin use. Literature evidence of liver disease being associated with metformin-associated metabolic acidosis is largely represented by case reports.

A recent study from Korea shows that in patients with type-2 diabetes mellitus, the mean FIB-4 score increased from 1.38 to 1.51 (p=0.001) after 2 years of metformin therapy, whereas the mean HSI score fell from 27.3 to 26.5 (p=0.001).

While these studies established that hepatic fat and pancreatic volume are high even in non-obese patients with T2DM, we were unable to estimate of hepatic and pancreatic fat precisely due to non-availability of advanced fat-imaging MRI software.

Review of Literature: Effects of SGLT2 Inhibitors and Abdominal Adipose Tissue Depots Metformin is an effective agent which helps to achieve better blood glucose control. This drug also benefits in the reduction of weight and blood pressure. Metformin results in weight loss.

Effect on Fat Mass:

Apart from weight loss, Metformin has been shown to reduce fat. It was reported that the use of Metformin significantly reduces body weight in T2DM patients on metformin therapy and inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

Overweight & obese (BMI 23.0 -35 kg/m2) subjects aged 30-60 years with T2DM of less than 5 year duration with HbA1c 6.5% to 9% & on a stable dose of metformin and/or sulphonylureas over last 8 weeks, fatty liver on ultrasound.

Exclusion Criteria:

The sample patient excluded in this study who had following medical history like: hypoglycaemia, diabetic abscess/ulcers, ketoacidosis, pregnant or lactating women, women planning for pregnancy/gestational diabetes, severe cardiac and renal disease, patients with renal transplant /undergoing immunosuppressive therapy for renal transplant ,substantial alcohol consumption, Child-Pugh B/C cirrhosis, other causes of liver disease, confounding concomitant drug use (including insulin, incretin mimetics, thiazolidinediones, vitamin E), and disorders such as a medical history of pancreatitis, pancreatic lipomatosis or pancreatic calculi (as detected by ultrasonography) ,type 1 diabetes mellitus.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To assess the effect of metformin on Pancreatic fat and hepatic fat in T2DM patients. | 120 days
  T2DM patients will undergo MRI, Ultrasound and Fibroscan testing to determine the level of fat in pancreas and liver.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Fortis CDOC Hospital
Locations (1):
- Anoop misra, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No